CLINICAL TRIAL: NCT00432549
Title: Evaluation of Almotriptan and Topiramate in the Detoxification and Treatment of Subjects With Medication Overuse Headache
Brief Title: Detoxification and Treatment of Subjects With Medication Overuse Headache
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The New England Center for Headache, P.C. (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAPSS-328
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2007-02-08 (Estimated); Status verified 2007-02

CONDITIONS: Analgesic Rebound Headache
Keywords: Medication overuse
MeSH Terms: conditions — Headache Disorders, Secondary; Prescription Drug Overuse | interventions — almotriptan; Topiramate

INTERVENTIONS:
Drug: Almotriptan
Drug: Topiramate

SUMMARY:
The purpose of this study is to assess the benefits of almotriptan used as a transitional therapy and topiramate in subjects with medication overuse headaches (MOH.

ELIGIBILITY:
Inclusion Criteria:

* Medication overuse headaches 18 years of age and older Must have a diagnosis of probable medication overuse headache Must have greater than fifteen headache days per month Must be in generally good health Female subjects must be postmenopausal or practicing an acceptable method of birth control

Exclusion Criteria:

* Not overusing six or more tablets per day of compounds containing barbituates opioids No overuse of triptans Previous failure or side effects with topiramate or almotriptan Cannot be pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-01; Study Completion 2007-02

PRIMARY OUTCOMES:
Primary measure for the detoxification period
Number of days with mild or no pain in the first two weeks of treatment
Primary for the prevention of relapse
Pain free days through day ninety

SECONDARY OUTCOMES:
Primary measure for the detoxification period
Number of days without any headache in the first two weeks of treatment
Primary for the prevention of relapse
Headache frequency through day ninety

CONTACTS AND LOCATIONS:
Overall Officials: Fred D Sheftell, M.D., Principal Investigator — The New England Center for Headache, P.C.
Locations (1):
- The New England Center for Headache, P.C., Stamford, Connecticut, United States